CLINICAL TRIAL: NCT06368921
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Biodistribution Characteristics, Biological Effects and Initial Efficacy of Recombinant Oncolytic Virus M1 for Injection (VRT106) in the Treatment of Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of Recombinant Oncolytic Virus M1(VRT106) in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-C01
Record Dates: First submitted 2024-04-09; First posted 2024-04-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRT106 (Experimental): VRT106
  Interventions: Biological: VRT106

INTERVENTIONS:
Biological: VRT106 — intratumoral injection

SUMMARY:
To Evaluate the safety and tolerability of single and multiple intratumoral injections of recombinant oncolytic virus M1 (VRT106) in patients with locally advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open-label, dose-escalation clinical study which aims to evaluate the safety and tolerability of IT injections of VRT106 in subjects with locally advanced/metastatic solid tumors, as well as evaluating the biological distribution characteristics and biological effects of VRT106 (i.e., virus tissue distribution and shedding characteristics), evaluating immunogenicity of VRT106, and preliminarily exploring the anti-tumor effects of VRT106.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an Institutional Review Board -approved informed consent prior to performing any of the Screening Visit procedures.
* Males and females at 18-75 years of age, inclusive, at the Screening Visit.
* Subjects must have histological or cytological diagnosis of locally advanced or metastatic solid tumors who are intolerable or refractory to the standard therapy.
* Have at least one injectable lesion.
* An Eastern Cooperative Oncology Group (ECOG) score of 0-1.
* An estimated survival time of ≥ 12 weeks.

Exclusion Criteria:

* Subject has received any anti-tumor treatment 4 weeks before using the IMP.
* Subject has received any prior oncolytic viruses or other gene therapies.
* Subject has a history of primary or acquired immunodeficient states, leukemia, lymphoma, acquired immunodeficiency syndrome (AIDS) or other clinical manifestations of infection with human immunodeficiency viruses, and those on immunosuppressive therapy.
* Subject has received immunomodulatory drugs, including but not limited to thymosin, IL-2, IFN, etc. within 14 days prior to first administration of IMP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of intratumoral injection of VRT106. | About 2 years
  Incidence rate of TEAE
Characterize the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) levels. | About 2 years
  Incidence rate of DLT

SECONDARY OUTCOMES:
Examine the biological distribution characteristics and shedding patterns of intratumoral injection of VRT106. | About 2 years
  Measure the distribution and shedding of VRT106 following intratumoral injection using qPCR (quantitative polymerase chain reaction) method.
Assess the immunogenicity of intratumoral injection of VRT106. | About 2 years
  Detect the presence of neutralizing antibodies against VRT106, which represent the potency of the neutralizing antibodies, using the PD50 value.
Assess the anti-tumor effect of VRT106, including objective response rate (ORR) as efficacy indicators. | About 2 years
  ORR is defined as the proportion of participants who have a partial response (PR) or complete response (CR) to intervention, based on assessments by RECIST v1.1.
Assess the anti-tumor effect of VRT106, including disease control rate (DCR) as efficacy indicators. | About 2 years
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) based on assessments by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No